CLINICAL TRIAL: NCT00217763
Title: A Phase III Study of the Efficacy and Safety of 3APS as Add-on Therapy in Mild to Moderate Alzheimer's Disease
Brief Title: European Study of 3APS in Mild to Moderate Alzheimer's Disease Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bellus Health Inc. - a GSK company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: CL-758010
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2007-12-10 (Estimated); Status verified 2007-12

CONDITIONS: Alzheimer's Disease
Keywords: Dementia; Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease; Dementia

INTERVENTIONS:
Drug: 3APS

SUMMARY:
The purpose of this Phase 3 study is to evaluate the efficacy and safety of 3APS as an add-on therapy to most standard medication for Alzheimer's disease compared to placebo (inactive substance pill) in patients with mild to moderate Alzheimer's disease.

DETAILED DESCRIPTION:
* Duration of treatment: 18 months
* 3 treatment arms:

Placebo and 2 different doses of active drug.

ELIGIBILITY:
RECRUITMENT OF PARTICIPANTS IS PERFORMED ONLY BY STUDY SITES.

INCLUSION CRITERIA:

Participants must meet the following inclusion criteria to be eligible.

* Male or Female (age 50 years and older): Female must be of non-childbearing potential (i.e. surgically sterilized or at least 2 years post-menopausal).
* Diagnosis of probable Alzheimer's disease based on the National Institute of Neurological and Communicative Disorders and Stroke/Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA criteria).
* Severity of dementia of mild to moderate degree as assessed by the Mini Mental State Examination (MMSE) performed at the screening visit.
* Patient must be living in the community with a reliable caregiver. Participant living in an assisted living facility may be included if study medication intake is supervised and participant has a reliable caregiver.
* Potential participant must be treated with an acetylcholinesterase inhibitor (donepezil, galantamine or rivastigmine) and must be on stable dose for at least 4 months prior to the screening visit and during the entire study period.
* Participants must not have taken memantine for at least 4 months prior to the commencement of screening. The use of memantine is prohibited during the course of the study.
* Fluency (oral and written) in the language in which the standardized tests will be administered.
* Signed informed consent from potential participant or legal representative and caregiver.

EXCLUSION CRITERIA:

Patients will not be eligible to participate in the study if they meet any of the following criteria:

* Potential participant with any other cause of dementia.
* Life expectancy less than 2 years.
* Potential participant with a clinically significant and/or uncontrolled condition or other significant medical disease.
* Previous use of anti-amyloid or vaccine treatment for Alzheimer's disease.
* Use of an investigational drug within 30 days prior to the screening visit or during the entire study.
* Previous exposure to 3APS.
* Inability to swallow pills.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 930 (Estimated)
Dates: Start 2005-09; Study Completion 2007-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Pr. Bruno Vellas, Principal Investigator — University Hospital Center, Toulouse
Locations (69):
- Belgium (4):
  - Middelheim Ziekenhuis Lindendreef, Antwerp
  - University Hospital Antwerp - Neurology - Prof. Dr. Patrick Cras, MD, PhD, Edegem
  - Memory Clinic University Hospital Gasthuisberg, Neurology Department, Leuven
  - Memory Centre, Polycliniques Brull, CHU de Liège, Liège
- France (12):
  - Besançon
  - Hôpital Pellegrin CHU de Bordeaux, Bordeaux
  - Dijon
  - Centre Hospitalier Régional Universitaire de Lille, Lille
  - Hôpital Sainte Marguerite Service de neuro-geriatrie, Marseille
  - Hôpital Gui de Chauliac - Service de Neurologie du Pr J. Touchon, Montpellier
  - Centre Mémoire de Ressources et de Recherche Hôpital Pasteur, Nice
  - Hôpital BROCA, Paris
  - CHU Reims- Hôpital Sébastopol-Service de médecine interne et Gérontologie Clinique, Reims
  - Hôpital Hôtel Dieu - Consultation de Gérontologie, Rennes
  - CHU Purpan, Toulouse
  - Tours
- Germany (8):
  - Charité Campus Benjamin Franklin - Universitätsmedizin Berlin - Klinik und Hochschulambulanz für Psychiatrie und Psychotherapie, Berlin
  - Johann-Wolfgang Goethe-Universität - Klinik für Psychiatrie und Psychotherapie, Frankfurt
  - Klinik für Psychiatrie und Psychotherapie - University Hospital Hamburg-Eppendorf - Dept. of Psychiatry and Psychotherapy, Hamburg
  - Psychiatrische Universitätsklinik Heidelberg - Sektion für Gerontopsychiatrie - Gedächtnisambulanz, Heidelberg
  - Gemeinschaftspraxis, Langendreer
  - Arzneimittelforschung Leipzig GmbH, Leipzig
  - Abteilung für Geriatrische Psychiatrie - Zentralinstitut für seelische Gesundheit - Universität Heidelberg, Mannheim
  - Munich
- Italy (8):
  - IRCCS Centro San Giovanni di Dio- Fatebenefratelli, Brescia
  - San Martino Hospital - Padiglione Specialita' Fondi, Genova
  - Dept. of Neurosciences TCR - University of Modena and Reggio Emilia, Modena
  - Perugia
  - Department of Neuroscience - Section of Neurology - University of Pisa, Pisa
  - Universita' Cattolica del Sacro Cuore, Rome
  - Rome
  - Vicenza
- Netherlands (4):
  - Medisch Centrum Alkmaar, Alkmaar
  - Dept. of Neurology and Alzheimer Center - Vrije Universiteit Medical Center, Amsterdam
  - Blaricum
  - Memory Clinic UMC St Radboud - Alzheimer Centre, Nijmegen
- Poland (6):
  - Bydgoszcz
  - Krakow
  - Lodz
  - Sopot
  - Warsaw
  - Wroclaw
- Spain (9):
  - Barakaldo
  - Fundaciò ACE- Institut Català de Neurociències Aplicades, Barcelona
  - Hospital del Mar- Servicio de Neurologia, Barcelona
  - Hospital Santa Creu i Sant Pau, Servicio de Neurología, Unitad de Memoria, Barcelona
  - Unitat de Valoració de la Memòria i les Demències - Hospital Santa Caterina - Institut d'Assistència Sanitària, Girona
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitairo La Paz, Madrid
  - Hospital Universitario Ramón y Cajal - Unidad de Geriatria, Madrid
  - Pamplona
- Sweden (7):
  - Linköping
  - Lund
  - Neuropsychiatric Clinic - University Hospital MAS, Malmo
  - Mölndal
  - Enheten för klinisk Läkemedelsforskning - Minnesmottagningen - Karolinska Universitetssjukhuset - Huddinge, Stockholm
  - Memory clinic - Uddevalla Hospital, Uddevalla
  - Memory Clinic -Geriatric Centre - Academic Hospital, Uppsala
- Switzerland (2):
  - Memory Clinic - Neuropsychology Center - University Hospital, Basel
  - Geneva
- United Kingdom (9):
  - Research Institute for Care of Elderly - St Martin's Hospital, Bath
  - Fylde Medical Clinic, Blackpool
  - Memory Assessment Centre, Blackpool
  - Wales College of Medicine - Llandough Hospital, Cardiff
  - East Sussex
  - Glasgow Memory Clinic - Golden Jubilee National Hospital, Glasgow
  - Murray Royal Hospital, Perth
  - Memory Assessment Centre - Moorgreen Hospital, Southampton
  - Kingshill Research Centre - Victoria Hospital, Swindon

REFERENCES:
- See also: Related Info — http://www.neurochem.com